CLINICAL TRIAL: NCT02986399
Title: Influence of a Fast Track Pathway for Hip Fracture Patients on Mortality and Quality of Life
Brief Title: Fast Track Hip Fracture - an Optimized Pathway for Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Other Study IDs: 284907
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Hip Fractures
Keywords: fast track
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard care: Hip fracture patients operated at Akershus University hospital in 2012 and 2013.
- Fast track patient pathway: Hip fracture patients operated at Akershus University hospital in 2014 and 2015.
  Interventions: Other: Fast track patient pathway

INTERVENTIONS:
Other: Fast track patient pathway — Admittance: Ambulance - Radiology - Orthopaedic ward. Focus on preoperative information, stress reduction, pain relief, early mobilization and nutritional status.
  Groups: Fast track patient pathway

SUMMARY:
The study examines if the introduction of a fast track pathway for hip fracture patients had an influence on mortality and quality of life by comparing these outcomes between all hip fracture patients operated at Akershus University Hospital two years before and two years after this change in standard care.

DETAILED DESCRIPTION:
The Norwegian hip fracture register prospectively collects data on all hip fracture patients including, among others, time to surgery, type of fracture, type of surgery and American Society of Anesthesiologists (ASA) score. The register also collects quality of life data 4 and 12 months after surgery. Using the unique Norwegian personal identification number the data from the Norwegian hip fracture register will be connected with data from the electronic patient record at Akershus University hospital (AHUS). Fast track surgery for hip fracture patients was introduced at the end of 2013. Mortality and quality of life data will be compared for all hip fracture patients operated at AHUS two years before and two years after this change in standard care. The combined data from the register and the electronic patient records will be used for regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Operated at Akershus university hospital for a hip fracture (neck of femur, trochanteric, subtrochanteric) in 2012, 2013, 2014 or 2015
* 18 years or older

Exclusion Criteria:

* stress fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hip fracture patients operated at Akershus university hospital in 2012, 2013, 2014 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 2495 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
30 day mortality rate | Within 30 days from surgery
  Percentage of patients who die within 30 days from hip fracture surgery

SECONDARY OUTCOMES:
1 year mortality rate | Within 1 year from surgery
  Percentage of patients who die within 1 year from hip fracture surgery
Quality of life | 4 and 12 months from surgery
  Quality of life measured by EQ-5D
Readmissions | Within 30 days from discharge
  Unscheduled, all-cause readmission within 30 days from discharge from the index admission
Postoperative infection | Within 1 year from surgery
  Superficial and / or deep surgical site infection
Re-operation | Within 1 year from surgery
  All-cause re-operation at the site of the index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Asbjorn Aaroen, Professor, Study Director — Akershus University Hospital and Faculty of Medicine, University of Oslo

IPD SHARING:
Plan to Share IPD: No